CLINICAL TRIAL: NCT06498908
Title: Success Rate of Intracervical Balloon Placement With Nitrous Oxide Administration. A Randomized Control Study
Brief Title: Intracervical Balloon Placement With Nitrous Oxide Administration
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Scott Chudnoff, Dr. Scott Chudnoff, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N20A
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Labor Pain; Induced; Birth
Keywords: pregnancy
MeSH Terms: conditions — Labor Pain | interventions — Nitrous Oxide; Oxygen

STUDY DESIGN:
Intervention Model Description: Nitrous Oxide vs Oxygen
Who Masked: Participant
Masking Description: Subjects won't be told which group they were assigned. Care providers will be told which group subject is assigned/
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrous Oxide (Experimental): Patients in the intervention arm will receive an inhalant of 50% nitrous/50% oxygen intended to target pain relief for the duration of their foley ballon placement.
  Interventions: Drug: Nitrous oxide
- Oxygen (Placebo Comparator): Patients in the control arm will receive an inhalant of 100% oxygen for the duration of their foley balloon placement.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Nitrous oxide — Nitrous oxide, commonly known as laughing gas, is a colorless, non-flammable gas with a slightly sweet odor, used for its analgesic and anesthetic properties in medical and dental procedures to provide pain relief and sedation.
  Arms: Nitrous Oxide
Drug: Oxygen — Oxygen is a colorless, odorless gas essential for human respiration and used medically to treat conditions resulting from low oxygen levels in the blood. In this trial Oxygen is being used as a placebo.
  Arms: Oxygen

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of nitrous oxide versus oxygen in facilitating the successful placement of a Foley balloon catheter for cervical ripening and induction of labor.

DETAILED DESCRIPTION:
This is a single center randomized controlled trial aimed to compare the effectiveness of nitrous oxide versus oxygen in facilitating the successful placement of a Foley balloon catheter for cervical ripening and induction of labor. Pregnant women requiring labor induction will be randomly assigned to receive either nitrous oxide or oxygen during the Foley balloon placement. The primary outcome measured will be the success rate of the Foley balloon placement, with secondary outcomes including patient comfort, pain levels during the procedure, and any adverse effects. The study seeks to determine if nitrous oxide can improve the success rate of Foley balloon placement compared to oxygen and to evaluate the overall patient experience and safety associated with its use in this context.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to labor and delivery for induction of labor (term inductions, medically indicated preterm inductions).
* Pregnant patients who are eligible for intracervical balloon placement.

Exclusion Criteria:

* Pregnant patients with contraindications to receiving nitrous oxide.
* Inability to safely self-administer nitrous oxide
* Allergy to nitrous oxide
* History of malignant hyperthermia,
* Concomitant administration of magnesium sulfate
* Less than 35 weeks gestational age
* Non-reassuring fetal heart tracing
* Use of intravenous or intramuscular opioid within 4 hours
* Vitamin B12 deficiency
* Gas-trapping conditions such as pneumothorax or small bowel obstruction
* Patients requesting neuraxial anesthesia
* Non-English speaking patients.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
success rate of intracervical balloon placement | 15 minutes
  successfull placement of intracervical ripening ballon on first attempt

SECONDARY OUTCOMES:
Pain Relief | 15 minutes
  Patients reported a pain score of a three or less for the duration of the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Maimonides Medical Center OB/GYN, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No